CLINICAL TRIAL: NCT07387237
Title: Multigene Germline Panel Testing in Gastric Cancer Patients in Portugal
Status: Completed | Type: Observational
Sponsor: Unidade Local De Saúde Do Norte Alentejano (Other)
Responsible Party: Principal Investigator, Beatriz Mourato, MD, Unidade Local De Saúde Do Norte Alentejano
Other Study IDs: MGPT Gastric Cancer; MGPT Gastric Cancer (Other: 1)
Record Dates: First submitted 2025-10-01; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer (Diagnosis); Stomach Cancer
Keywords: Multigene Germeline Panel Test; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multigene germeline panel test in gastric cancer patients

DETAILED DESCRIPTION:
We conducted a retrospective observational study including 51 patients with histologically confirmed gastric cancer who underwent MGPT between 2020 and 2025. Genetic testing was performed using validated 15 or 30 gene panels. Clinical, pathological, and survival data were retrieved from medical records.

ELIGIBILITY:
Inclusion Criteria

* Eligible participants were adults (≥18 years) with histologically confirmed gastric adenocarcinoma who underwent MGPT between 2020 and 2025;
* Ability to understand Portuguese and/or English;
* Ability to provide valid informed consent.

Exclusion Criteria:

* All patients who met eligibility and inclusion criteria were included in the study;
* Patients without a definitive genetic report or with incomplete clinical data for key study variables were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with histologically confirmed gastric adenocarcinoma who underwent MGPT between 2020 and 2025
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
MGPT result | 5 years
  positive vs negative

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade Local de Saúde do Alto Alentejo, Portalegre, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT07387237/Prot_SAP_000.pdf
  • Informed Consent Form: Inform Const Form (2024-09-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT07387237/ICF_001.pdf